CLINICAL TRIAL: NCT03224728
Title: Effect of Spherical Aberration on the Optical Quality After Implantation of Two Different Aspherical Intraocular Lenses
Brief Title: Spherical Aberration on the Optical of Two Different Aspherical Intraocular Lenses
Status: Completed | Type: Observational
Sponsor: Hospital Hietzing (Other)
Responsible Party: Principal Investigator, Michael Lasta, Principal investigator, Hospital Hietzing
Other Study IDs: EK-12-256-0113
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 2 different Intraocular lenses: 2 different intraocular lenses were compared
  Interventions: Device: intraocular lens

INTERVENTIONS:
Device: intraocular lens

SUMMARY:
Purpose: To compare the effect of spherical aberration on optical quality in eyes with two different aspherical intraocular lenses Methods: In this prospective, randomized clinical trial 120 eyes of 60 patients underwent phacoemulsification. In patient's eyes an aberration-free aspherical IOL (Aspira-aA; Human Optics) or an aberration-correcting aspherical IOL (Tecnis ZCB00; Abott Medical Optics) were randomly implanted. Three months after surgery visual acuity, contrast sensitivity, wavefront measurements with iTrace as well as tilt and decentration measurements with Visante anterior segment OCT were performed.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral age-related cataract
* Potential postoperative visual acuity of 1.0 Snellen
* No relevant ocular pathology other than cataract
* Written informed consent to surgery and participation in the study

Exclusion Criteria:

* Amblyopia, diabetic retinopathy, uveitis or other relevant ophthalmic diseases
* Optical media disturbances due to: corneal and vitreal opacity, PEX
* Preceding ocular trauma or ocular surgery within 6 months
* Inability to cooperate
* Pregnancy (a pregnancy test will be performed preoperatively in women of reproductive age)

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men and women between 50 and 85 years with age related cataract
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Modulation transfer function (MTF) at 3 months after surgery | 3 months

REFERENCES:
- [Derived] Lasta M, Mihaltz K, Kovacs I, Vecsei-Marlovits PV. Effect of Spherical Aberration on the Optical Quality after Implantation of Two Different Aspherical Intraocular Lenses. J Ophthalmol. 2017;2017:8039719. doi: 10.1155/2017/8039719. Epub 2017 Aug 16. PMID 28900544